CLINICAL TRIAL: NCT07102576
Title: A Phase 1, Open-Label Study to Assess Psychological and Biological Effects of MDMA Assisted Therapy When Administered to Mental Health Providers in Training to be MDMA-Assisted Therapists
Brief Title: MDMA-Assisted Therapy for Mental Healthcare Providers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rachel Yehuda (Other)
Responsible Party: Sponsor-Investigator, Rachel Yehuda, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY-24-00412
Record Dates: First submitted 2025-07-31; First posted 2025-08-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Mental Wellbeing
Keywords: Psychedelic Therapy; MDMA; MDMA-Assisted Therapy; Mental Health; Therapist
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-Label (Experimental): One session of MDMA-Assisted Therapy
  Interventions: Drug: MDMA Hydrochloride

INTERVENTIONS:
Drug: MDMA Hydrochloride — Initial dose of 120 mg MDMA HCl in a therapeutic setting, followed 1.5 to 2 hours later by a supplemental dose of 40 mg MDMA HCl. Supplemental doses may be withheld if tolerability issues emerge or it is declined by the participant.

SUMMARY:
This is a phase 1, open-label study to assess changes in mental well-being following MDMA administration within a therapeutic setting, in mental health providers who are in training to become MDMA assisted therapists. Secondary outcome measures will examine the effects on provider burnout, provider self-efficacy, mood, self-compassion, quality of life, and other psychological factors. Participants will work with a co-therapy pair as they engage in a preparatory session, one experimental session with MDMA, and an integration session the following day.

DETAILED DESCRIPTION:
This study is investigating the psychological and biological effects and safety of MDMA-assisted therapy (MDMA-AT) in healthy volunteers who are: 1) mental healthcare providers or trainees, and 2) learning or have been certified to conduct MDMA-AT. As research in MDMA-AT expands, there is a need to evaluate the safety and efficacy of MDMA-assisted therapy in healthy volunteers, in order to better understand its effects in populations beyond clinical samples and to inform future comparisons. This study will assess whether a relatively brief intervention (consisting of one MDMA-AT session with one preparatory and one integration session) can improve overall mental wellbeing in a healthy sample of mental healthcare providers, while also evaluating its effects on provider burnout, self-assessed counselor efficacy, mood, psychological flexibility, quality of life, and experiential avoidance. In addition, this study supports continued training for new MDMA-AT providers, including the option for their own MDMA experience to expand on their knowledge of the subjective effects and therapeutic potential of MDMA-AT and enhance their qualifications to provide that therapy. Participants will engage in structured preparation, treatment, and follow-up, guided by trained clinical professionals. Assessments will take place throughout the study to monitor mental health outcomes and ensure participant well-being. Participation will consist of: - Screening Period (up to 4 weeks): Phone screen, informed consent, eligibility assessment, and enrollment. - Preparatory Period (1-4 weeks): Preparatory session with study clinicians, baseline assessments. - Treatment Period (2 days): Experimental session (MDMA administered in a controlled therapeutic setting) followed by an integrative session the next day. - Follow-Up Period (up to 4 weeks): Follow-up visit approximately one month after experimental session, outcome assessments, and study termination.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years at the time of signing the informed consent.
* Fluent in English
* Able to swallow pills
* Agree to have study visits audiovisually recorded
* Able to provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of the participant becoming unwell or unreachable.
* Must be licensed, license-eligible, or trainees in a relevant healthcare/mental health profession
* Must be learning or have been certified to conduct MDMA-assisted therapy through the Lykos MDMA-Assisted Therapy Training program or authorized affiliate program
* Body weight of at least 45 kilograms (kg; or 100 pounds (lbs)).

Exclusion Criteria

* Have engaged in a new form of psychiatric or mental health care within 12 weeks of enrollment
* Have a current alcohol or cannabis use disorder of any severity within the 12 months prior to enrollment
* Have a substance use disorder of any severity within 12 months prior to enrollment
* Any suicidal ideation within the last 6 months
* Repetitive or recent use of Ecstasy/MDMA
* Current enrollment in any other clinical study involving an investigational study treatment or any other type of medical research, unless approved by the study clinician
* Meet diagnostic criteria for a Major Depressive Episode currently or within the prior 3 months or meet diagnostic criteria for a current anxiety disorder assessed
* Have a current eating disorder with compensatory behaviors
* Have a history of, or a current primary psychotic disorder or bipolar disorder
* Previous participation in a clinical trial that included administration of MDMA
* Individuals in a personal relationship with the site investigator
* Are pregnant or nursing or are able to become pregnant and are not practicing an effective means of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-09-21 (Estimated); Study Completion 2029-12-21 (Estimated)

PRIMARY OUTCOMES:
Mental Health Continuum-Short Form (MHC-SF) | At baseline and 28 days post-treatment
  The MHC-SF is a self-report measure consisting of 14 questions rated for the frequency at which they are experienced, on a scale from "0-never" to "5-every day" within the past month. The MHC-SF is a shortened version of the Mental Health Continuum Long Form (MHC-LF), a 40-item measure which was developed to assess emotional, social, and psychological well-being, a three factor structure validated in national and international populations. The MHC-SF was developed using a subset of items from the MHC-LF to represent each of these three well-being constructs: The MHC-SF yields a total score range of 0-70, where higher scores reflect greater mental well-being. Subscale ranges are: Emotional Well-Being: 0-15 (3 items), Psychological Well-Being: : 0-30 (6 items), and Social Well-Being: 0-25 (5 items). Subscale scores reflect functioning in each domain, while the total score captures overall mental well-being.

SECONDARY OUTCOMES:
The Maslach Burnout Inventory - Human Services Survey (MBI-HSS) | At baseline and 28 days post-treatment
  The MBI-HSS is a 22-item survey scored from 0-6 per item, producing a total score range of 0-132, where higher scores indicate poorer health outcomes. This 22-item survey addresses 3 scales: Emotional Exhaustion: 0-42, which measures feelings of being emotionally overextended and exhausted by one's work; Depersonalization: 0-42, which measures an unfeeling and impersonal response toward recipients of one's service, care treatment, or instruction; and Personal Accomplishment: 0-48, which measures feelings of competence and successful achievement in one's work.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Glatman Zaretsky, Study Director — Mount Sinai Icahn School of Medicine; Rachel Yehuda, Principal Investigator — Mount Sinai Icahn School of Medicine
Locations (1):
- The Parsons Research Center for Psychedelic Healing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plans at this time